CLINICAL TRIAL: NCT03825718
Title: A Study of GC007F CAR-T Cell Immunotherapy for Relapsed or Refractory B- ALL
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hebei Yanda Ludaopei Hospital (Other)
Collaborators: Gracell Biotechnology Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PGC0002
Record Dates: First submitted 2019-01-22; First posted 2019-01-31 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2019-01

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T treatment group (Experimental): The patients will receive one dose of GC007F. GC007F dosage ranges from 6×10^4 to 2×10^6 CAR+T/Kg.
  Interventions: Biological: GC007F

INTERVENTIONS:
Biological: GC007F — GC007F is the CAR-T cell immunotherapy targeted CD19. The subjects will receive GC007F as one dose. The dosage ranges from 6×10^4 to 2×10^6 CAR+T/Kg.

SUMMARY:
The study is an early, open, single-centered trial.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the safety and tolerance of GC007F CAR-T cell immunotherapy in relapsed or refractory B-ALL. The study will include 20 subjects to receive GC007F therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory paediatric B-cell ALL 1) 2nd or greater bone marrow (BM) relapse or 2) Relapse after remission for the first time in 12 months or 3) The interval between relapse after allogeneic hematopoietic stem cell transplantation and CAR-T cells transfusion≥100 days or 4) Primary refractory as defined by not achieving a CR after 2 cycles of a standard chemotherapy regimen or chemorefractory as defined by not achieving a CR after 1 cycle of standard chemotherapy for relapsed leukaemia or 5) Patients with Philadelphia chromosome positive ALL were eligible if they were intolerant to or had failed two lines of tyrosine kinase inhibitor (TKI) therapy, or if TKI therapy was contraindicated or 6) Ineligible for allogeneic SCT because of: i. Comorbid disease ii. Other contraindications to allogeneic SCT conditioning regimen iii. Lack of suitable donor iv. Prior SCT v. Declined allogeneic SCT as a therapeutic option after documented discussion, including expected outcomes, about the role of SCT with a BM transplantation physician not part of the study team
2. For relapsed patients, CD19 tumour expression demonstrated in bone marrow or peripheral blood by flow cytometry within 3 months of study entry
3. Aged 2-70 years
4. Eastern cooperative oncology group (ECOG) performance status of 0 to 2
5. Life expectancy≥12 weeks
6. Adequate organ function defined as:1) Creatinine clearance (as estimated by Cockcroft Gault) >60 mL/min. 2) Serum ALT/AST<2.5 ULN. 3) Total bilirubin<1.5 mg/dl, except in subjects with Gilbert's syndrome. 4) Cardiac ejection fraction≥45%, no evidence of pericardial effusion as determined by an ECHO, and no clinically significant ECG findings. 5) No clinically significant pleural effusion. 6) Baseline oxygen saturation >92% on room air. 7) pulmonary function: ventilation function is normal or is restricted mildly.
7. Females of reproductive age must be in non-lactation period. Females of childbearing potential must have a negative serum or urine pregnancy test. All subjects must use medical-approved-contraception (such as intrauterine device and contraceptive drugs) during the period of trial and in 6 months after cell transfusion therapy.
8. The subject agree to and sign informed consent form, willing and able to comply with the planned visit, research, treatment planning, laboratory and other test procedures.

Exclusion Criteria:

1. Isolated extra-medullary disease relapse;
2. Patients with Burkitt's lymphoma/leukaemia;
3. Central nervous system leukemia involved CNS3;
4. Concomitant malignancy other than non-melanoma skin cancer or adequately-treated cervical carcinoma in situ or prostate cancer (PSA score<1.0) or adequately-treated low grade bladder cancer or surgery-cured ductal carcinoma in situ or diagnosis of other malignancy exceeds 5 years without relapse or treatment during the 5 years;
5. Concomitant genetic diseases except Down syndrome;
6. Any result of the following virology tests is positive: HIV; HCV; HBsAg; or HBCAb positive with HBV DNA copies positive(≥ 5×10^2 copies/ml); RPR+TPPA postive;
7. Live vaccine ≤4 weeks prior to apheresis;
8. Prior CD19 targeted therapy with the exception of subjects who received GC007F in this study and are eligible for re-treatment; Prior chimeric antigen receptor therapy or other genetically modified T cell therapy;
9. Presence of grade 2 to 4 graft-versus-host disease (GVHD) after allo-HSCT;
10. The following medications were excluded: 1) Steroids: Therapeutic systemic doses of steroids must be stopped >72 hours prior to tisagenlecleucel infusion. However, the following physiological replacement doses of steroids are allowed: <12 mg/m^2/day hydrocortisone or equivalent; 2) Allogeneic cellular therapy: Any donor lymphocyte infusions must be completed >6 weeks prior to cell infusion; 3) GVHD therapies: Any systemic drug used for GVHD must be stopped >4 weeks prior to infusion to confirm that GVHD recurrence is not observed;
11. Prior treatments of CNS diseases must be stoped >3 days prior to infusion (e.g., intrathecal injection of methotrexate) 1) Radiotherapy of non-CNS nidus must be completed >2 weeks prior to infusion; 2) CNS stereotactic radiotherapy must be completed >8 weeks prior to infusion;
12. ≥2 grade toxicities related to previous therapy are not relieved, with the exception of adverse events without safety risk (e.g., alopecia);
13. Known life-threatening allergy, hypersensitivity or intolerance to GC007F cells and adjuvant, including DMSO (see investigator's brochure);
14. Patients with active autoimmune disease (e.g., systemic lupus erythematosus, sjogren syndrome, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease) receive immunosuppressive therapy in 4 weeks before inclusion. thyroid hormone replacement therapy is an exception;
15. For patients that underwent major surgical operation before CAR-T treatment, or anticipated to undergo a major surgical operation during the study process, they need to be fully recovered and clinically stable before inclusion.
16. Participate in other clinical trial and received study drugs <28 days prior to inclusion;
17. Concomitant disease that may or severe medical condition that may affect patients' safety, including active viral or bacterial infection, uncontrollable systemic fungal infection, uncontrollable cardiac disease, hypertension, abuse of psychoactive drugs, et al.
18. Any other condition that may increase subjects' risk or interfere with trial's results.

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Dose Limiting Toxicity | 12 weeks
  A dose limiting toxicity is defined as any toxicity that is considered to be primarily related to the GC007F cells, which is irreversible, or life threatening or hematologic or non-hematologic Grade 3-5
Incidence and severity of adverse events | 12 weeks
  After GC007F infusion, adverse events will be graded as CTCAE 4.0
GC007F persistence | 12 weeks
  After GC007F infusion, GC007F CAR copies in peripheral blood. bone marrow and CSF will be measured by qPCR in 12 weeks

SECONDARY OUTCOMES:
Percents of Patients with best response as complete remission and MRD negative complete remission. | 12 weeks
  Response rates will be estimated as the percents of patients whose best response is complete remission and MRD negative complete remission.

CONTACTS AND LOCATIONS:
Overall Officials: Peihua Lu, MD/PHD, Principal Investigator — HeiBei YanDa Ludaopei hospital
Locations (1):
- Hebei Yanda Ludaopei Hospital, Sanhe, Hebei, China